CLINICAL TRIAL: NCT05494047
Title: A Phase III, Randomized, Double-blind and Controlled Clinical Trial to Evaluate the Immunogenicity and Safety of Influenza Vaccine, Inactivated, Quadrivalent Developed by Sinovac Biotech Co., Ltd. Compared to a Licensed Quadrivalent Influenza Vaccine, VaxigripTetra™, in Individuals Aged 3 Years and Older in Chile
Brief Title: Phase Ⅲ, Clinical Trial to Compare an Inactivated Quadrivalent Influenza Vaccine and a Licensed Vaccine in Chile
Acronym: TetraFluVac
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Sinovac Biotech (Chile) SpA (Industry); Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-QINF-3004
Record Dates: First submitted 2022-08-07; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Influenza; Vaccines
Keywords: influenza; vaccine; immunogenicity; clinical-trial
MeSH Terms: conditions — Influenza, Human | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Individuals will be randomized to receive Vaxigrip Tetrs TM or equivalent vaccine developed by Sinovac Biotech Co. It is a a comparative, double blind, propsective clinical trial with 2 active compunds.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomized by a computer system. Investigators and care providers will not be able to know the vaccine administered. Statistical analysis will not have access to the information of immunization. Nonetheless, personnel study who will administer the vaccine will know the group because they will have access to the envelope of the vaccine then this personnel will not have any other responsibility during the study moreover, they will not have mantain regular contact with investigational team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tetravalent influenza vaccine developed by Sinovac Biotech Co. (Experimental): The group will be formed by 800 individuals. 200 from 3 to 8 years old, 200 from 9 to 17 years old, 200 from 18 to 64 years old and 200 subjects 65 years and older. They will receive an unique dose of the tetravalent influenza vaccine developed by Sinovac Biotech Co.(H1N1, H3N2 and 2 strains of influenza B). Subjects 3 to 8 years will receive 2 doses of influenza vaccine unless they have receipt of 2 previous doses of any influenza vaccine or they have an history of previous influenza.
  Interventions: Drug: Tetravalent influenza vaccine developed by Sinovac Biotech Co.
- Vaxigrip Tetra TM (Active Comparator): The group will be formed by 800 individuals. 200 from 3 to 8 years old, 200 from 9 to 17 years old, 200 from 18 to 64 years old and 200 subjects 65 years and older. They will receive an unique dose of the tetravalent influenza vaccine Vaxigrip Tetra TM(H1N1, H3N2 and 2 strains of influenza B). Subjects 3 to 8 years will receive 2 doses of influenza vaccine unless they have receipt of 2 previous doses of any influenza vaccine or they have an history of previous influenza.
  Interventions: Drug: Tetravalent influenza vaccine developed by Sinovac Biotech Co.

INTERVENTIONS:
Drug: Tetravalent influenza vaccine developed by Sinovac Biotech Co. — 15μg Hemagglutinin Antigen (HA) of each of the four strains
  Other Names: Sinovac vaccine

SUMMARY:
This study compares the immunogenity and safety of quadrivalent inactivated influenza vaccines. The experimental group receives the quadrivalent influenza vaccine developed by Sinovac Biotech Co., Ltd and the control group immunized with Vaxigrip Tetra™. The group has 1600 persons from general population 3 years and older. The design is double-blind and randomized. The primary outcome is the immunogenicity against the 4 strains of influenza included in both vaccines.

DETAILED DESCRIPTION:
The study is designed to evaluate the immunogenicity of the quadrivalent inactivated-virus influenza vaccine developed by Sinovac Biotech Co., Ltd against Vaxigrip Tetra™. The population included in the study is healthy subjects 3 years and older, being 800 individuals 10 years old or less and 800 over 18 years, randomized 1:1 to experimental vaccine or Vaxigrip Tetra™. Volunteers 8 years old or less, without history of previous influenza infection will receive 2 doses of vaccine, al other individuals will receipt 1 dose of vaccine. Immunogenicity will be assessed one month after the last dose of vaccine, humoral responses will be determined for all patients meanwhile ome subgroup of patients will have a determination of cellular immunity also. Subjects will be follow up for one month, adverse events will be assessed during this time.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers age 3 years and older, in good health or medically stable;
2. Written informed consent obtained from subjects or/and legal guardian;
3. No receipt of influenza vaccines within 6 months or plans to receive any influenza vaccines during the study;
4. Female subjects of non-childbearing may be enrolled in the study. Nonchildbearing potential is defined as surgically sterile (history of bilateral tubal ligation, bilateral oophorectomy, hysterectomy) or premenarche or postmenopausal (defined as amenorrhea for ≥ 12 consecutive months prior to screening without an alternative medical cause).
5. Female subjects of childbearing potential may be enrolled in the study, if the subject:

   * Has a negative pregnancy test on the day of the first dose (day 0);
   * Has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first dose and until at least 28 days after vaccination.

Exclusion Criteria:

1. History of seasonal influenza within 6 months prior to the study entry;
2. Axillary temperature ≥37.3℃;
3. History of Guillain-Barré syndrome within 6 weeks of receipt of prior influenza vaccine.
4. History of allergy to any vaccine, or any ingredient of the experimental vaccine.
5. Serious adverse reaction(s) to the vaccine, such as urticaria, dyspnea or angioneurotic edema, etc.;
6. History of serious neurological disorder (such as epilepsy, convulsions, etc.) , or mental illness;
7. Autoimmune disease or immunodeficiency/immunosuppressive, or any immunosuppressant receipt within 6 months prior to the study entry;
8. Significant chronic illnesses that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion (may include, but are not limited to cardiovascular disease, hypertension and diabetes that cannot be controlled by drugs, liver or kidney disorders, HIV infection or malignant tumor;
9. Acute central nervous system diseases such as encephalitis/myelitis, acute disseminating encephalomyelitis, and related disorders;
10. Absence of spleen, functional absence of spleen, and absence or removal of spleen under any circumstances;
11. Diagnosed coagulation function abnormal (e.g., coagulation factor deficiency, coagulation disorder, or platelet abnormalities), or obvious bruising or coagulation disorders;
12. Alcoholism or history of drug abuse
13. Acute disease or acute stage of chronic disease within 7 days prior to study entry;
14. Received blood products within 3 months prior to study entry;
15. Received any live attenuated vaccine within 14 days prior to study entry or any subunit vaccine or inactivated vaccine within 7 days prior to study entry;
16. Pregnant women or lactating women;
17. Subjects participate other clinical trials (licensed or unlicensed vaccines, drugs, organisms, devices, blood products or drugs) during the study period;
18. Any other factors which are unsuitable for participation in the clinical trial as judged by the investigator.

    -

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Seroconversion for influenza | 28 days after the last dose of vaccination
  Seroconversion rates and geometric mean titers of human influenza antibody for each of the four antigens.

SECONDARY OUTCOMES:
Antibody titer 1:40 or more | 28 days after the last dose of vaccination
  Proportion of subjects with antibody titer ≥1:40
Cellular immunity-ELISPOT | 28 days after the last dose
  Quantification by ELISPOT of specific Spot Forming Cells for cytokines, molecules and immunoglobulins induced by both vaccines
Cellular immunity-Cytometry | 28 days after the last dose
  Quantification by flow cytometry of CD3+CD4+ and CD3+CD8+ cells positive for Activation Induced Markers, induced by both vaccines.
Cellular immunity-Luminex (TM) | 28 days after the last dose
  • Quantification by Luminex® of cytokines secreted by specific CD3+CD4+ and CD3+CD8+ cells induced by each vaccine

OTHER OUTCOMES:
Adverse events (AEs) | Solicited AEs within 7 days after each dose and unsolicited AEs within 28 days after each dose
  Local and systemic AEs
Serious adverse events | Within 28 days after each dose
  Ocurrence and relationship of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Pablo A Gonzalez, PhD, Principal Investigator — Pontifical Catholic University of Chile
Locations (5):
- Chile (5):
  - Hospital Puerto Montt, Port Montt, Los Lagos Region
  - Centro de Investigaciones Médicas Respiratorias (CIMER), Providencia, Santiago Metropolitan
  - Hospital Clínico UC Christus, Santiago, Santiago Metropolitan
  - Hospital Félix Bulnes, Santiago, Santiago Metropolitan
  - Clínica Alemana de Santiago, Vitacura, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaccines against influenza WHO position paper - November 2012. Wkly Epidemiol Rec. 2012 Nov 23;87(47):461-76. No abstract available. English, French. PMID 23210147
- [Background] Reed C, Meltzer MI, Finelli L, Fiore A. Public health impact of including two lineages of influenza B in a quadrivalent seasonal influenza vaccine. Vaccine. 2012 Mar 2;30(11):1993-8. doi: 10.1016/j.vaccine.2011.12.098. Epub 2012 Jan 5. PMID 22226861
- [Background] Lee BY, Bartsch SM, Willig AM. The economic value of a quadrivalent versus trivalent influenza vaccine. Vaccine. 2012 Dec 14;30(52):7443-6. doi: 10.1016/j.vaccine.2012.10.025. Epub 2012 Oct 19. PMID 23084849
- [Background] Jain VK, Domachowske JB, Wang L, Ofori-Anyinam O, Rodriguez-Weber MA, Leonardi ML, Klein NP, Schlichter G, Jeanfreau R, Haney BL, Chu L, Harris JS, Sarpong KO, Micucio AC, Soni J, Chandrasekaran V, Li P, Innis BL. Time to Change Dosing of Inactivated Quadrivalent Influenza Vaccine in Young Children: Evidence From a Phase III, Randomized, Controlled Trial. J Pediatric Infect Dis Soc. 2017 Mar 1;6(1):9-19. doi: 10.1093/jpids/piw068. PMID 28062552
- [Background] Cadorna-Carlos JB, Nolan T, Borja-Tabora CF, Santos J, Montalban MC, de Looze FJ, Eizenberg P, Hall S, Dupuy M, Hutagalung Y, Pepin S, Saville M. Safety, immunogenicity, and lot-to-lot consistency of a quadrivalent inactivated influenza vaccine in children, adolescents, and adults: A randomized, controlled, phase III trial. Vaccine. 2015 May 15;33(21):2485-92. doi: 10.1016/j.vaccine.2015.03.065. Epub 2015 Apr 2. PMID 25843270
- [Background] Mallory RM, Yu J, Kameo S, Tanaka M, Rito K, Itoh Y, Dubovsky F. The safety and efficacy of quadrivalent live attenuated influenza vaccine in Japanese children aged 2-18 years: Results of two phase 3 studies. Influenza Other Respir Viruses. 2018 Jul;12(4):438-445. doi: 10.1111/irv.12555. Epub 2018 Apr 10. PMID 29573143
- [Background] Claeys C, Drame M, Garcia-Sicilia J, Zaman K, Carmona A, Tran PM, Miranda M, Martinon-Torres F, Thollot F, Horn M, Schwarz TF, Behre U, Merino JM, Sadowska-Krawczenko I, Szymanski H, Schu P, Neumeier E, Li P, Jain VK, Innis BL. Assessment of an optimized manufacturing process for inactivated quadrivalent influenza vaccine: a phase III, randomized, double-blind, safety and immunogenicity study in children and adults. BMC Infect Dis. 2018 Apr 18;18(1):186. doi: 10.1186/s12879-018-3079-8. PMID 29669531
- [Background] Beran J, Peeters M, Dewe W, Raupachova J, Hobzova L, Devaster JM. Immunogenicity and safety of quadrivalent versus trivalent inactivated influenza vaccine: a randomized, controlled trial in adults. BMC Infect Dis. 2013 May 20;13:224. doi: 10.1186/1471-2334-13-224. PMID 23688546
- [Background] Greenberg DP, Robertson CA, Noss MJ, Blatter MM, Biedenbender R, Decker MD. Safety and immunogenicity of a quadrivalent inactivated influenza vaccine compared to licensed trivalent inactivated influenza vaccines in adults. Vaccine. 2013 Jan 21;31(5):770-6. doi: 10.1016/j.vaccine.2012.11.074. Epub 2012 Dec 8. PMID 23228813